CLINICAL TRIAL: NCT06102057
Title: PACCELIO - FDG-PET Based Small Volume Accelerated Immuno Chemoradiotherapy in Locally Advanced NSCLC
Acronym: PACCELIO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: TheraOp (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESR-21-21536; 2022-003408-33 (EudraCT Number); ARO 2023-06 (Other: ARO)
Record Dates: First submitted 2023-09-08; First posted 2023-10-26 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Stage III Non-small Cell Lung Cancer; Locally Advanced; Unresectable
Keywords: chemoradiotherapy; immunotherapy; small volume accelerated chemoradiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy; Immunotherapy

STUDY DESIGN:
Intervention Model Description: Experimental Arm (FDG-PET-based small volume accelerated radiotherapy with concurrent standard of care chemotherapy) Conventional Arm (standard FDG-PET-based radiotherapy with concurrent standard of care chemotherapy)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Arm (Active Comparator): standard FDG-PET-based radiotherapy with concurrent standard of care chemotherapy
  Interventions: Radiation: standard Radiotherapy; Drug: Chemotherapy; Drug: Immunotherapy
- Experimental Arm (Experimental): FDG-PET-based small volume accelerated radiotherapy with concurrent standard of care chemotherapy
  Interventions: Drug: Chemotherapy; Drug: Immunotherapy; Radiation: Experimental Radiotherapy

INTERVENTIONS:
Radiation: standard Radiotherapy — standard FDG-PET-based radiotherapy
  Other Names: standard
  Arms: Conventional Arm
Drug: Chemotherapy — concurrent standard of care chemotherapy
  Other Names: standard
Drug: Immunotherapy — standard of care consolidation therapy with durvalumab (fixed dose of 1500 mg q4w) for up to 12 months or until progression of disease, unacceptable toxicity, patient´s wish, or investigator´s decision, whichever comes first.
  Other Names: standard
Radiation: Experimental Radiotherapy — FDG-PET-based small volume accelerated radiotherapy
  Other Names: Experimental
  Arms: Experimental Arm

SUMMARY:
Multinational, randomized, controlled, open-label, multicenter phase II trial. Eligible patients will be randomized in a ratio of 1:1 to Experimental Arm (FDG-PET-based small volume accelerated radiotherapy with concurrent standard of care chemotherapy) or Conventional Arm (standard FDG-PET-based radiotherapy with concurrent standard of care chemotherapy). Patients showing complete response, partial response, or stable disease following chemoradiotherapy will receive standard of care consolidation therapy with durvalumab (fixed dose of 1500 mg q4w) for up to 12 months or until progression of disease, unacceptable toxicity, patient´s wish, or investigator´s decision, whichever comes first.

After end of durvalumab therapy, patients will undergo safety follow up for 90 (+7) days followed by survival follow up until overall end of study. Overall end of study will be reached 24 months after the last patient has started durvalumab therapy. Patients showing PD following chemoradiotherapy will be treated according to investigator´s decision but will be followed up until overall end of study.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Patients irrespective of sex and gender, aged 18 years or older at the time of signing the ICF
* Patients must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the study as determined by the investigator
* Patients with histologically or cytologically documented NSCLC who present with locally advanced, unresectable (Stage III) disease (according to version 8 of the International Association for the Study of Lung Cancer Staging Manual in Thoracic Oncology (IASLC Staging Manual in Thoracic Oncology 2016))
* Patients fit for simultaneous chemoradiotherapy and consolidation immunotherapy according to interdisciplinary consensus
* Histologically proven PD-L1-expression of ≥ 1% (tumor proportion score; TPS) in tumor sample as assessed in routine staging using a validated test such as Ventana SP236 assay
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1 at enrolment
* Tumor assessment by FDG-PET CT within 21 days prior to start of chemoradiotherapy.
* Adequate pulmonary function test results

  * Pre- or post-bronchodilator forced expiratory volume 1 of 1.0 L or >40% of predicted AND
  * Diffusing capacity of the lung for carbon monoxide (DLCO) >30% of predicted
* Adequate bone marrow and organ function at enrolment

  * Hemoglobin ≥9.0 g/dL
  * Absolute neutrophil count >1.5 × 109/L
  * Platelet count >100 × 109/L
  * Serum bilirubin ≤1.5 × upper limit of normal (ULN)
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 × ULN
  * Measured creatinine clearance (CrCl) >40 mL/min or calculated CL >40 mL/min as determined by Cockcroft-Gault (using actual body weight)
* Body weight of >30 kg at enrolment
* Evidence of post-menopausal status, or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they are amenorrhoic for 12 months or more without an alternative medical cause. The following age-specific requirements apply:

  * Women <50 years old would be considered post-menopausal if they have been amenorrhoic for 12 months or more following cessation of exogenous hormonal treatments with luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution
  * Women ≥50 years old would be considered post-menopausal if they have been amenorrhoic for 12 months or more following cessation of all exogenous hormonal treatments, radiation-induced oophorectomy with last menses >1 year ago, chemotherapy-induced menopause with >1 year interval since last menses, or surgical sterilization (bilateral oophorectomy or hysterectomy)
* Women of childbearing potential (WOCBP) and male patients with partners of childbearing potential must agree to always use a highly effective form of contraception according to the Clinical Trials Facilitation and Coordination Group during the treatment phase of this study and for at least 90 days after the last dose durvalumab or 6 months after the last dose of chemotherapy, whichever occurs last

Exclusion Criteria:

* Mixed small cell and NSCLC histology
* Neuroendocrine tumor
* Distant metastases
* Malignant pleural effusion or pericardial effusion
* Acute superior vena cava obstruction
* Receipt of prior or current cancer treatment for NSCLC, including but not limited to, surgical resection, radiation therapy, investigational agents, chemotherapy, and monoclonal antibodies (mAbs). Exception: Prior surgical resection of limited metachronous NSCLC (i.e., stage I or II) is permitted.
* Receipt of live attenuated vaccine within 30 days prior to the start of therapy. Note: Patients, if enrolled, should not receive live vaccine during treatment phase and up to 30 days end of treatment
* Major surgical procedure (as defined by the Investigator) within 28 days prior start of treatment.
* Prior exposure to immune-mediated therapy, including but not limited to, other anti-CTLA-4, anti-PD-1, anti-PD-L1 (including durvalumab), and anti-PD-L2 antibodies, including therapeutic anticancer vaccines
* Current use of ongoing long-term immunosuppressive medication. The following are exceptions to this criterion

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
* History of allogeneic organ transplantation
* Active or prior documented autoimmune or inflammatory disorders including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia
  * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Patients without active disease in the last 5 years at randomization may be included but only after consultation with the local study physician
  * Patients with celiac disease controlled by diet alone
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, ILD, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs, or compromise the ability of the patient to give written informed consent
* Patients with oxygen dependence
* Acute inflammation of mediastinal lymph nodes/mediastinal lymphadenopathy in the context of active pneumoconiosis, sarcoidosis or tuberculosis
* History of another primary malignancy, except for

  * Basal cell carcinoma of the skin
  * Second malignancy diagnosed > 2 years prior to NSCLC diagnosis if after curative treatment without persistence or progression at baseline. Patients with a previous history of radiation therapy are eligible provided field overlap is minimal and the risk of toxicity to tissues in the overlapping region(s) is deemed to be acceptable by treating radiation oncologist.
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease
* History of leptomeningeal carcinomatosis
* Positive diagnostic test for hepatitis B (hepatitis B surface antigen) or hepatitis C (hepatitis C antibody or hepatitis C RNA)
* Known active infection of tuberculosis or human immunodeficiency virus
* Known allergy or hypersensitivity to concomitant chemotherapy and durvalumab or any of the excipients
* Any medical contraindication to treatment with platinum-based doublet chemotherapy as listed in the applying SmPCs
* Patients who have disease considered for surgical treatment as part of their care plan, such as Pancoast or superior sulcus tumors.
* Concurrent enrolment in another clinical study, unless it is an observational (noninterventional) clinical study or the follow-up period of an interventional study
* Participation in another clinical study with an investigational product during the 4 weeks prior to enrolment
* Pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Comparison of the Completion rate of Experimental Arm to Conventional Arm | approximately 22 weeks after start of radio-chemotherapy
  To assess the feasibility of an FDG-PET-based small volume accelerated chemoradiotherapy followed by immunotherapy with durvalumab compared to standard FDG-PET-based chemoradiotherapy followed by immunotherapy with durvalumab Completion rate defined as rate of patients having received:
  * the prescribed radiotherapy dose ± 2 fractions and
  * simultaneous platinum-based chemotherapy and · immunotherapy consolidation with durvalumab starting within 42 days after the last dose of chemoradiotherapy and
  * either at least 3 doses of durvalumab or less than 3 doses of durvalumab in case immunotherapy was permanently discontinued due to documented extrathoracic immune-related toxicity.

SECONDARY OUTCOMES:
Comparison of the Occurrence of adverse events and serious events of Experimental Arm to Conventional Arm | up to 78 weeks
  To assess the safety and tolerability of an FDGPET- based small volume accelerated chemoradiotherapy followed by immunotherapy with durvalumab compared to standard FDG-PET-based chemoradiotherapy followed by immunotherapy with durvalumab
  Occurrence of adverse events and serious events:
  * adverse events grade ≥ 3 (according to NCI CTCAE v5.0)
  * SAEs
  * Unexpected AEs
Comparison of the Time to locoregional progression of Experimental Arm to Conventional Arm | time from randomization to progression in the primary tumor or any of mediastinal lymph nodes, up to 143,5 weeks
  Assess efficacy of FDG-PET-based smallvolumeaccelerated CRT followed by immunotherapy compared to standard FDG-PET-based CRT followed by immunotherapy in terms of time to locoreg. progression, time to locoreg. in- and out-of-RTfield progress
  - Time to locoregional progression
Comparison of the Time to locoregional in-RT-field progression of Experimental Arm to Conventional Arm | time from rando to progression in primary tumor or mediastinal lymph nodes within the target volume, up to 143,5 weeks
  Assess efficacy of FDG-PET-based smallvolumeaccelerated CRT followed by immunotherapy compared to standard FDG-PET-based CRT followed by immunotherapy in terms of time to locoreg. progression, time to locoreg. in- and out-of-RTfield progress
  · Time to locoregional in-RT-field progression
Comparison of the Time to locoregional out-of-RT-field progression of Experimental Arm to Conventional Arm | time from rando to progression in mediastinal lymph nodes outside the target volume, up to 143,5 weeks
  Assess efficacy of FDG-PET-based smallvolumeaccelerated CRT followed by immunotherapy compared to standard FDG-PET-based CRT followed by immunotherapy in terms of time to locoreg. progression, time to locoreg. in- and out-of-RTfield progress
  · Time to locoregional out-of-RT-field progression
Comparison of the Time to distant progression time from rando to appearance of metastases elsewhere of Experimental Arm to Conventional Arm | time from rando to appearance of metastases elsewhere, up to 143,5 weeks
  Assess efficacy of FDG-PET-based smallvolumeaccelerated CRT followed by immunotherapy compared to standard FDG-PET-based CRT followed by immunotherapy in terms of time to locoreg. progression, time to locoreg. in- and out-of-RTfield progress
  · Time to distant progression time from rando to appearance of metastases elsewhere
Comparison of the PFS of Experimental Arm to Conventional Arm | time from rando to disease progression or death by any cause, up to 143,5 weeks
  Assess efficacy of FDG-PET-based smallvolumeaccelerated CRT followed by immunotherapy compared to standard FDG-PET-based CRT followed by immunotherapy in terms of time to locoreg. progression, time to locoreg. in- and out-of-RTfield progress
  · PFS
Comparison of the OS of Experimental Arm to Conventional Arm | time from rando to death by any cause, up to 143,5 weeks
  Assess efficacy of FDG-PET-based smallvolumeaccelerated CRT followed by immunotherapy compared to standard FDG-PET-based CRT followed by immunotherapy in terms of time to locoreg. progression, time to locoreg. in- and out-of-RTfield progress
  · OS
Comparison of the ORR of Experimental Arm to Conventional Arm | Objective response rate defined as the proportion of randomized patients with best response of complete or partial response, up to 143,5 weeks
  Assess efficacy of FDG-PET-based smallvolumeaccelerated CRT followed by immunotherapy compared to standard FDG-PET-based CRT followed by immunotherapy in terms of time to locoreg. progression, time to locoreg. in- and out-of-RTfield progress
  · ORR
Comparison of the DCR of Experimental Arm to Conventional Arm | Disease control rate defined as the proportion of rando patients with best response of complete response, partial response, or stable disease, up to 143,5 weeks
  Assess efficacy of FDG-PET-based smallvolumeaccelerated CRT followed by immunotherapy compared to standard FDG-PET-based CRT followed by immunotherapy in terms of time to locoreg. progression, time to locoreg. in- and out-of-RTfield progress
  · DCR
Comparison of the Change in symptoms of Experimental Arm to Conventional Arm | up to 143,5 weeks
  Assess symptoms and patient-reported QoL in patients receiving an FDG-PET-based smallvolumeaccelerated CRT followed by immunotherapy compared to patients receiving standard FDG-PET-based CRT followed by immunotherapy
  1. Change in symptoms assessed with the EORTC QLQ-C30
  2. Change in symptoms assessed with the EORTC QLQ-LC13
  The results of the questionnaire are usually presented as scale scores, ranging from 0 to 100. Higher scores on the symptom scales indicate a worse quality of life.
Comparison of the Change in functioning of Experimental Arm to Conventional Arm | up to 143,5 weeks
  Assess symptoms and patient-reported QoL in patients receiving an FDG-PET-based smallvolumeaccelerated CRT followed by immunotherapy compared to patients receiving standard FDG-PET-based CRT followed by immunotherapy
  1. Change in functioning assessed with the EORTC QLQ-C30
  2. Change in functioning assessed with the EORTC QLQ-LC13
  The results of the questionnaire are usually presented as scale scores, ranging from 0 to 100. Higher scores on the functional scales indicate a better quality of life.
Comparison of the Change in global health-status/QoL of Experimental Arm to Conventional Arm | up to 143,5 weeks
  Assess symptoms and patient-reported QoL in patients receiving an FDG-PET-based smallvolumeaccelerated CRT followed by immunotherapy compared to patients receiving standard FDG-PET-based CRT followed by immunotherapy
  1. Change in global health-status/QoL assessed with the EORTC QLQ-C30
  2. Change in global health-status/QoL assessed with the EORTC QLQ-LC13
  The results of the questionnaire are usually presented as scale scores, ranging from 0 to 100. Higher scores on the global health and quality of life scale indicate a better quality of life.
To assure radiotherapy quality in terms of percentage of patients without major protocol deviations of ≥85% | up to 55 months
  Percentage of patients without major protocol deviations regarding radiotherapy quality

OTHER OUTCOMES:
To exploratively analyze the impact of lesional FDG uptake in baseline PET/CT as predictive factor for response to radio-chemo-immunotherapy, PFS, and survival | time from randomization to disease progression or death by any cause, up to 143,5 weeks
  Quantifiable imaging parameters (e.g., SUV) will be correlated to response and survival outcomes, reflected in separate protocol to be setup
  SUV is a common unitless measurement for radioactivity uptake. In the study we will measure maximum SUV and mean SUV from tumor volume. The tumor volume with the unit millilitre will be measured by an automatic segmentation were any area with SUV above a threshold value of 40% of SUVmax will be attributed to the tumor volume. These imaging parameters will be correlated with time to progression from randomization
To exploratively analyze anatomic (RECIST)/metabolic (PERCIST) response to chemoradiotherapy in FDG-PET/CT at the end of chemoradiotherapy as predictive factor for overall response, response to consolidating immunotherapy, PFS, and survival | time from randomization to disease progression or death by any cause, up to 143,5 weeks
  Quantifiable imaging parameters (e.g., SUV) will be correlated to response and survival outcomes, reflected in separate protocol to be setup
  SUV is a common unitless measurement for radioactivity uptake. In the study we will measure maximum SUV and mean SUV from tumor volume. The tumor volume with the unit millilitre will be measured by an automatic segmentation were any area with SUV above a threshold value of 40% of SUVmax will be attributed to the tumor volume. These parameters will be correlated with time to progression from randomization Also, for changes of measurements of SUVmax and SUVmax from baseline correlation will be done with time to progression. In this analyisis also changes in tumor diameter (measured from CT) and changes in tumor volume (measured from PET) will be included into the analysis.
Exploratively evaluate add.effect of consolidation immunotherapy measured 3 months after the end of CRT on metabolic response beyond that measured at the end of CRT, further PFS and survival as potential hint for necessary treatment intensification | time from randomization to disease progression or death by any cause, up to 143,5 weeks
  Quantifiable imaging parameters (e.g., SUV) will be correlated to response and survival outcomes, reflected in separate protocol to be setup
  SUV is a common unitless measurement for radioactivity uptake. In the study we will measure maximum SUV and mean SUV from tumor volume. The tumor volume with the unit millilitre will be measured by an automatic segmentation were any area with SUV above a threshold value of 40% of SUVmax will be attributed to the tumor volume. These imaging parameters will be correlated with time to progression from randomization Further changes of measurements of SUVmax, SUVmax, tumor diameter and tumor volume from end of chemoradiation therapy will be correlated with time to progression in the subgroup receiving three PET/CT scans.
To exploratively analyze the impact of the neutrophil to lymphocyte ratio (NLR) as predictive biomarker for response to consolidating immunotherapy and survival | up to 55 months
  Relation of NLR to response and survival outcomes, reflected in separate protocol to be setup
  It is calculated by dividing the number of neutrophils by number of lymphocytes.
To exploratively analyze the impact of the ALI Index as predictive biomarker for response to consolidating immunotherapy and survival | up to 55 months
  Relation of ALI Index (Advance lung cancer inflammation) to response and survival outcomes, reflected in separate protocol to be setup
  ALI is calculated as (BMI x Alb / NLR) where BMI = body mass index, Alb = serum albumin, NLR (neutrophil lymphocyte ratio, a marker of systemic inflammation).
To exploratively analyze the effective radiotherapy dose to immune cells (EDIC) as predictive factor for immunocompetence | up to 55 months
  Relation of EDIC to immunomarkers (NLR), reflected in separate protocol to be setup
  The EDIC model considers the exposure of circulating immune cells as the proportion of blood flow to lung, heart, liver, and the volume of the exposed area of the body, with the basis of mean lung dose, mean heart dose, mean liver dose and integral dose of the body region which are to be extracted from the RT plan. EDIC will be calculated as described in Xu et al. 2020.
  NLR is calculated by dividing the number of neutrophils by number of lymphocytes.
To exploratively analyze the effective radiotherapy dose to immune cells (EDIC) as predictive factor for immunocompetence | up to 55 months
  Relation of EDIC to immunomarkers (ALI), reflected in separate protocol to be setup
  The EDIC model considers the exposure of circulating immune cells as the proportion of blood flow to lung, heart, liver, and the volume of the exposed area of the body, with the basis of mean lung dose, mean heart dose, mean liver dose and integral dose of the body region which are to be extracted from the RT plan. EDIC will be calculated as described in Xu et al. 2020.
  ALI is calculated as (BMI x Alb / NLR) where BMI = body mass index, Alb = serum albumin, NLR (neutrophil lymphocyte ratio, a marker of systemic inflammation).
To exploratively analyze the effective radiotherapy dose to immune cells (EDIC) as predictive factor for response to chemoradio-immunotherapy | up to 55 months
  Relation of EDIC to response to chemoradio-immunotherapy, reflected in separate protocol to be setup
  The EDIC model considers the exposure of circulating immune cells as the proportion of blood flow to lung, heart, liver, and the volume of the exposed area of the body, with the basis of mean lung dose, mean heart dose, mean liver dose and integral dose of the body region which are to be extracted from the RT plan. EDIC will be calculated as described in Xu et al. 2020.
To exploratively analyze the effective radiotherapy dose to immune cells (EDIC) as predictive factor for survival. | up to 55 months
  Relation of EDIC to survival outcomes, reflected in separate protocol to be setup
  The EDIC model considers the exposure of circulating immune cells as the proportion of blood flow to lung, heart, liver, and the volume of the exposed area of the body, with the basis of mean lung dose, mean heart dose, mean liver dose and integral dose of the body region which are to be extracted from the RT plan. EDIC will be calculated as described in Xu et al. 2020.

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Nestle, Prof., Principal Investigator — Kliniken Maria Hilf GmbH; Stefan Rieken, Prof., Principal Investigator — Universitätsmedizin Göttingen (UMG)
Locations (11):
- Germany (10):
  - Universitätsklinik Carl Gustav Carus der Technischen Universität Dresden, Dresden
  - Universitätsklinikum Essen - Klinik für Strahlentherapie, Essen
  - Medical Center - University Of Freiburg, Department of Radiation Oncology, Freiburg im Breisgau
  - Universitätsmedizin Göttingen, Department for Radiotherapy and Radiooncology, Göttingen
  - Universität des Saarlandes, Klinik für Strahlentherapie und Radioonkologie, Homburg
  - Kliniken Maria Hilf GmbH Mönchengladbach, Mönchengladbach
  - Klinikum der Universitaet Muenchen AöR, Department of Radiotherapy and Radiation Oncology, München
  - Pius-Hospital Oldenburg, Hematology and Oncology, Oldenburg
  - Vinzenz Von Paul Kliniken gGmbH, Klinik für Strahlentherapie und Palliativmedizin, Stuttgart
  - Überörtliche Berufsausübungsgemeinschaft Troisdorf, Troisdorf
- Universitätsspital Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No